CLINICAL TRIAL: NCT03556410
Title: Sleep, Exercise and Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jill Kanaley, Professor, University of Missouri-Columbia
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Sleep and Exercise
Record Dates: First submitted 2018-05-23; First posted 2018-06-14 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Obesity
Keywords: Sleep; Obesity; Metabolic Syndrome; Physical Activity
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Motor Activity | interventions — Sleep; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sleep (Placebo Comparator): Subject will undergo 5 days of shortened sleep and then 2 days of ad libitum sleep.
  Interventions: Behavioral: sleep
- sleep+exercise (Experimental): Subject will undergo 5 days of shortened sleep but also have 45 min of moderate exercise/day and then 2 days of ad libitum sleep
  Interventions: Behavioral: sleep; Behavioral: exercise

INTERVENTIONS:
Behavioral: sleep — Shortened sleep will be requested of all subjects. During this time normal physical activity will be monitored.
Behavioral: exercise — Shortened sleep will be requested of all subjects. During this time normal physical activity will be monitored and 45 min of exercise will be required during the shortened sleep days .
  Arms: sleep+exercise

SUMMARY:
Insufficient or disrupted sleep, lack of physical activity and poor diet are linked with obesity and are now potential targets to combat obesity. Sleep related issues have become more important as people have been able to work, socialize, and use electronic devices outside of daylight hours. This has also altered how we eat and how we exercise. All of these factors can cause the body to not handle glucose (sugar) well resulting in insulin resistance. In time this could lead to type 2 diabetes.

DETAILED DESCRIPTION:
Experimental Design: Subjects will have preliminary screening tests. Two conditions (with/without exercise) will be completed in a randomized, crossover design. Subjects will wear an activity monitor (actigraph) and sleep monitor (actiwatch) for 14 days. For the first 7 days this is the lead in period for us to get baseline sleep day. For the following 5 days they will be asked to reduce their sleep with a specified bed time (ie. 11 pm - 5 am) followed by 2 days of ad libitum sleep hours, totaling 14 days for each condition. On one condition we will let them do their usual physical active and on the other condition during the shortened sleep they will be asked to exercise for 45 min each day at a moderate intensity (65% VO2max). Meal tests will be assessed after 7 days of normal habits, after 5 days of sleep deprivation, and after 2 days of ad libitum sleep, totaling 6 meal tolerance tests throughout the entirety of the study. Testing will be conducted at the MU Physical Activity and Wellness (MUPAW) center in Gwynn Hall and in McKee Gymnasium. Sleep logs will be done for 3 days prior to the meal test days and food diaries will be done 4 days prior.

Visit 1: Subjects will be provided a verbal explanation of the study and will sign the informed consent if interested. They will then complete questionnaires assessing health history, sleep, and physical activity habits. A DXA scan and anthropometrics will also be recorded. Participants will also perform a maximal peak oxygen consumption test (VO2max) on a treadmill for calculations during exercise regimen, 65% VO2max. A resting blood pressure will be measured three times with a sphygmomanometer. A mask will be securely fitted to the subject's face, covering the nose and mouth, and connected to the Parvo Medics TrueOne 2400 (Parvo Medics, Sandy, UT) metabolic cart via a flexible hose to monitor carbon dioxide expulsion and oxygen consumption. Heart rate will be monitored through a polar heart rate monitor chest strap (Polar Elctro, Kempele, Finland). Subjects will be sent home with a pulse oximeter to sleep with to ensure the subjects do not have sleep apnea.

Visit 2: Subjects will collect physical activity monitor (actigraph) and sleep monitor (actiwatch) along with surveys to fill out each day about dietary consumption, sleep habits and physical activity, lasting for 14 days.

Visit 3-5: Subjects will have their resting energy expenditure (REE) measured and then do a meal test. Subjects will arrive at MUPAW at ~7 am, following at least a 10 hour fast, abstain from caffeine for >10 hours and alcohol for 24 hours prior to arriving.

REE: A ParvoMedics TrueOne2400 metabolic measurement system (Sandy Lake, UT) will be used to measure REE. The REE measurement will occur in the morning after an overnight fast and after ingestion of the meal during testing. During the REE, participants will lay supine in a recliner for 30 min while all expired air is collected in a canopy that will be placed over the participants head and analyzed for O2 and CO2 content. The participants will be able to breath room air normally during the procedure. Expired air will be collected and the O2 and CO2 values in the expired air will be converted to a REE estimate using the ParvoMedics software.

Meal test: An IV catheter will be placed in a forearm vein (usually the antecubital vein). A mixed meal tolerance test will consist of a commercially available shake (16 ounces) that will be consumed within 10 minutes. Blood samples (~5 mL) will be collected over a 3 hour period from the start of the test meal ingestion.

Visit 6: Repeat of Visit 2.

Visit 7-9: Repeat of Visit 3-5. Exercise Sessions will be at McKee Gymnasium which will last 45 minutes for 5 days. A mask will be used to monitor oxygen consumption for 10 minutes at the start of the session to ensure appropriate work load.

Subjects will be reminded not to do any distance driving during their 5 days of shortened sleep.

2. Blinding, including justification for blinding or not blinding the trial. Describe un-blinding procedures.

Participants will be told at the beginning of the condition if they are going to be in the exercise condition or just being monitored for physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese men and women
* BMI of 25-35 kg/m2
* normally active (>5000 steps per day)
* normal sleeping habits of 7-9 hours per night

Exclusion Criteria:

* type 2 diabetics
* diagnosed with cardiovascular disease
* hypertensive
* smokers
* pregnant
* taking lipid-lowering medications
* have any recent changes in hormonal birth control
* night shift workers or take regular daytime naps
* on any medications known to impact metabolism, appetite, or sleep
* have any allergies to milk and soy
* sleep apnea or other sleep disorders
* if the 7 days of sleep monitoring prior to sleep restriction period shows inconsistent sleep hours outside of 7-9 hours per night.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
glucose tolerance | 3 hour glucose before the shortened sleep, 5 days after the shortened sleep and after 2 days of ad libitum sleep
  integrated area under the curve

SECONDARY OUTCOMES:
insulin | 3 hour insulin before the shortened sleep, 5 days after the shortened sleep and after 2 days of ad libitum sleep
  integrated area under the curve
FFA | fasting values at the beginning of the OGTT
  fasting FFA concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
We will share data on request that will be deidentified.